CLINICAL TRIAL: NCT01352676
Title: Validation of a Decision Rule to Limit CT Scanning in Suspected Renal Colic
Brief Title: Limit Computed Tomography (CT) Scanning in Suspected Renal Colic
Acronym: Prospective
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 1104008278; HS018322 (Other: Other Federal Funding)
Record Dates: First submitted 2011-05-10; First posted 2011-05-12 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Renal Colic; Flank Pain; Back Pain
Keywords: renal colic; flank pain; back pain
MeSH Terms: conditions — Renal Colic; Flank Pain; Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Computed tomography (CT) scanning is overused, expensive, and causes cancer. CT scan utilization in the U.S. has increased from an estimated 3 million CTs in 1980 to 62 million per year in 2007. From 2000 through 2006, Medicare spending on imaging more than doubled to $13.8 billion with advanced imaging such as CT scanning largely responsible. CT represents only 11% of radiologic examinations but is responsible for two-thirds of the ionizing radiation associated with medical imaging in the U.S. Recent estimates suggest that there will be 12.5 cancer deaths for every 10,000 CT scans. Renal colic is a common, non-life-threatening condition for which CT is overused. As many as 12% of people will have a kidney stone in their lifetime, and more than one million per year will present to the emergency department (ED). CT is now a first line test for renal colic, and is very accurate. However, 98% of kidney stones 5mm or smaller will pass spontaneously, and CT rarely alters management. A decision rule is needed to determine which patients with suspected renal colic require CT. While the signs and symptoms of renal colic have been shown to be predictable, no rule has yet been rigorously derived or validated to guide CT imaging in renal colic. A subset of patients with suspected renal colic may have a more serious diagnosis or a kidney stone that will require intervention; however the investigators maintain that clinical criteria, point of care ultrasound and plain radiography (when appropriate), will provide a more comparatively effective and safer approach by appropriately limiting imaging.

DETAILED DESCRIPTION:
Study Aim: The specific aim of this study is to prospectively validate the previously derived decision rule for obtaining a Flank Pain Protocol (FPP) CT scan in suspected renal colic.

The investigators will integrate the derived clinical decision rule from the ongoing retrospective analysis with gestalt clinician pre-test probability, point of care ultrasound, and plain radiography (when appropriate) to prospectively and observationally test the rule at two distinct clinical settings. CT results and 90-day follow-up will be used to determine predefined outcomes.

Study Hypothesis: Prospective observational testing of a clinical decision rule, combined with point of care ultrasound and plain radiography when appropriate, will categorize >85% of patients who will require intervention, validating a decision rule to avoid unnecessary CT.

This amendment comes from recent evidence and work at our institution to develop an "ultra-low dose" CT scan protocol (ULDCT) with an effective radiation dose close to that of a plain film of the abdomen (KUB), or near 1mSv (compared to 8.5mSv in current practice). While we expect the ULDCT to be better than a KUB at localizing and characterizing kidney stones, what is unknown is how the loss in resolution with an ultra-low dose CT protocol might affect this localization and characterization of stones relative to a regular dose CT (current protocol), as well as the ability to find alternate diagnoses. Incorporating this additional imaging study in a subgroup of patients during the observational phase will allow us to determine test characteristics of the ULDCT that will allow incorporation into the prospective phase. This will hopefully provide excellent evidence about how to implement an ultra-low dose CT scan in practice, ultimately leading to a dramatic reduction in radiation exposure for a large number of patients at Yale and other sites.

We filed an amendment 11-15-2011. This amendment comes from recent evidence and work at our institution to develop an "ultra-low dose" CT scan protocol (ULDCT) with an effective radiation dose close to that of a plain film of the abdomen (KUB), or near 1mSv (compared to 8.5mSv in current practice). While we expect the ULDCT to be better than a KUB at localizing and characterizing kidney stones, what is unknown is how the loss in resolution with an ultra-low dose CT protocol might affect this localization and characterization of stones relative to a regular dose CT (current protocol), as well as the ability to find alternate diagnoses. Incorporating this additional imaging study in a subgroup of patients during the observational phase will allow us to determine test characteristics of the ULDCT that will allow incorporation into the prospective phase. This will hopefully provide excellent evidence about how to implement an ultra-low dose CT scan in practice, ultimately leading to a dramatic reduction in radiation exposure for a large number of patients at Yale and other sites.

This amendment comes from recent evidence and work at our institution to develop an "ultra-low dose" CT scan protocol (ULDCT) with an effective radiation dose close to that of a plain film of the abdomen (KUB), or near 1mSv (compared to 8.5mSv in current practice). While we expect the ULDCT to be better than a KUB at localizing and characterizing kidney stones, what is unknown is how the loss in resolution with an ultra-low dose CT protocol might affect this localization and characterization of stones relative to a regular dose CT (current protocol), as well as the ability to find alternate diagnoses. Incorporating this additional imaging study in a subgroup of patients during the observational phase will allow us to determine test characteristics of the ULDCT that will allow incorporation into the prospective phase. This will hopefully provide excellent evidence about how to implement an ultra-low dose CT scan in practice, ultimately leading to a dramatic reduction in radiation exposure for a large number of patients at Yale and other sites.

Future Direction: Ultimately the investigators intend to implement the validated decision rule at both study sites to evaluate further the feasibility, physician acceptance and comparative effectiveness of our rule. Using standard dissemination techniques and integration of the rule into the computerized physician order entry (CPOE) system at our institutions the investigators will determine the actual reduction in the number of FPP CT scans ordered, clinical outcomes based on 90-day follow up, survey of physician acceptance of the rule as well as an comparative effective analysis. The investigators will submit an application at a later date nearing the end of our projected enrollment for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the adult YNHH ED and Shoreline Medical Center SMC ED who are

  * 18 years or older,
  * renal colic is suspected upon presentation to the ED suggested by flank pain, back pain, abdominal pain, and/or hematuria, and
  * the physician intends to order a CT FPP study for suspicion of a kidney stone. Members of all ethnic and racial groups are eligible.

Exclusion Criteria:

* Patients will be excluded for any one of the following reasons: patients that are

  * pregnant
  * prisoners
  * unable or unwilling to consent (including non-English speaking) and
  * with a history or physical evidence of recent trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population will be all patients aged 18 or above presenting to the Yale New Haven Hospital (YNHH) ED and Shoreline Medical Center (SMC) ED for whom a FPP CT scan is ordered by the treating physician for suspected renal colic. A total of 800-1000 patients will be enrolled over a 1.5 year period 6-2011 to 1-2013, matching the sex/race/ethnicity makeup of that found for the retrospective study.
  The population of the primary catchment area for YNHH is 350,000 and includes a diverse ethnic and cultural mix. Women and minorities are strongly represented in the population. Women represent approximately 51% of the ED population. The racial mix is approximately 50% White, not of Hispanic Origin; 33% Black, not of Hispanic Origin, 15% Hispanic; 1% Asian and 1% other. The ethnicity of SMC patients is mostly White and 54% female.
Sampling Method: Non-Probability Sample
Enrollment: 635 (Actual)
Dates: Start 2011-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Ultra Low Dose vs Regular CT Scans | Baseline-90 Days
  both the CT results and the follow-up documentation will be reviewed by two separate MD observers who are blinded to both the predictor variables and the outcome of the decision rule. CT results will be categorized as defined above, and intervention as defined above will either be considered present (immediate or delayed) or absent based on follow-up documentation. In the case where there is a discrepancy in the categorization of CT or intervention, a third reviewer will be used as a tie-breaker, with discussion amongst all parties to reach a consensus if this is not clear.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Moore, MD, Principal Investigator — Yale University School of Medicine, Emergency Medicine
Locations (2):
- United States (2):
  - Shoreline Medical Center, Guilford, Connecticut
  - Yale University, Emergency Department, New Haven, Connecticut

REFERENCES:
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Background] Brenner D, Elliston C, Hall E, Berdon W. Estimated risks of radiation-induced fatal cancer from pediatric CT. AJR Am J Roentgenol. 2001 Feb;176(2):289-96. doi: 10.2214/ajr.176.2.1760289. PMID 11159059
- [Background] Medicare Part B Imaging Services. General Accounting Office. Washington D.C., 2008.
- [Background] Mettler FA Jr, Wiest PW, Locken JA, Kelsey CA. CT scanning: patterns of use and dose. J Radiol Prot. 2000 Dec;20(4):353-9. doi: 10.1088/0952-4746/20/4/301. PMID 11140709
- [Background] Kalra MK, Maher MM, Toth TL, Hamberg LM, Blake MA, Shepard JA, Saini S. Strategies for CT radiation dose optimization. Radiology. 2004 Mar;230(3):619-28. doi: 10.1148/radiol.2303021726. Epub 2004 Jan 22. PMID 14739312
- [Background] Jindal G, Ramchandani P. Acute flank pain secondary to urolithiasis: radiologic evaluation and alternate diagnoses. Radiol Clin North Am. 2007 May;45(3):395-410, vii. doi: 10.1016/j.rcl.2007.04.001. PMID 17601499
- [Background] Fritzsche P, Amis ES Jr, Bigongiari LR, Bluth EI, Bush WH Jr, Choyke PL, Holder L, Newhouse JH, Sandler CM, Segal AJ, Resnick MI, Rutsky EA. Acute onset flank pain, suspicion of stone disease. American College of Radiology. ACR Appropriateness Criteria. Radiology. 2000 Jun;215 Suppl:683-6. No abstract available. PMID 11037484
- [Background] Teichman JM. Clinical practice. Acute renal colic from ureteral calculus. N Engl J Med. 2004 Feb 12;350(7):684-93. doi: 10.1056/NEJMcp030813. No abstract available. PMID 14960744
- [Background] Ripolles T, Errando J, Agramunt M, Martinez MJ. Ureteral colic: US versus CT. Abdom Imaging. 2004 Mar-Apr;29(2):263-6. doi: 10.1007/s00261-003-0098-7. No abstract available. PMID 15290956
- [Background] Catalano O, Nunziata A, Altei F, Siani A. Suspected ureteral colic: primary helical CT versus selective helical CT after unenhanced radiography and sonography. AJR Am J Roentgenol. 2002 Feb;178(2):379-87. doi: 10.2214/ajr.178.2.1780379. PMID 11804898
- [Background] Gottlieb RH, La TC, Erturk EN, Sotack JL, Voci SL, Holloway RG, Syed L, Mikityansky I, Tirkes AT, Elmarzouky R, Zwemer FL, Joseph JV, Davis D, DiGrazio WJ, Messing EM. CT in detecting urinary tract calculi: influence on patient imaging and clinical outcomes. Radiology. 2002 Nov;225(2):441-9. doi: 10.1148/radiol.2252020101. PMID 12409578
- [Background] Ripolles T, Agramunt M, Errando J, Martinez MJ, Coronel B, Morales M. Suspected ureteral colic: plain film and sonography vs unenhanced helical CT. A prospective study in 66 patients. Eur Radiol. 2004 Jan;14(1):129-36. doi: 10.1007/s00330-003-1924-6. Epub 2003 Jun 19. PMID 12819916
- [Background] Broder J, Bowen J, Lohr J, Babcock A, Yoon J. Cumulative CT exposures in emergency department patients evaluated for suspected renal colic. J Emerg Med. 2007 Aug;33(2):161-8. doi: 10.1016/j.jemermed.2006.12.035. Epub 2007 Jun 5. PMID 17692768
- [Background] Elton TJ, Roth CS, Berquist TH, Silverstein MD. A clinical prediction rule for the diagnosis of ureteral calculi in emergency departments. J Gen Intern Med. 1993 Feb;8(2):57-62. doi: 10.1007/BF02599984. PMID 8441076
- [Derived] Moore CL, Bomann S, Daniels B, Luty S, Molinaro A, Singh D, Gross CP. Derivation and validation of a clinical prediction rule for uncomplicated ureteral stone--the STONE score: retrospective and prospective observational cohort studies. BMJ. 2014 Mar 26;348:g2191. doi: 10.1136/bmj.g2191. PMID 24671981
- [Derived] Lukasiewicz A, Bhargavan-Chatfield M, Coombs L, Ghita M, Weinreb J, Gunabushanam G, Moore CL. Radiation dose index of renal colic protocol CT studies in the United States: a report from the American College of Radiology National Radiology Data Registry. Radiology. 2014 May;271(2):445-51. doi: 10.1148/radiol.14131601. Epub 2014 Jan 27. PMID 24484064